CLINICAL TRIAL: NCT00894075
Title: Single-Center, Case-Control Study of Safety, Efficacy and Pharmacokinetics of ENB-0040 (Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein) for Treatment of Hypophosphatasia in Children
Brief Title: Safety and Efficacy Study of ENB-0040 in Juvenile Patients With Hypophosphatasia (HPP)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn pending further review of clinical design.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-004-09
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Hypophosphatasia
Keywords: genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ENB-0040 — 1mg/kg subcutaneous injection thrice weekly for 6 months
  Other Names: Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein; sALP-Fc-D10

SUMMARY:
This Clinical Trial is being conducted to study Hypophosphatasia (HPP), a bone disorder caused by gene mutations or changes. These gene mutations cause low levels of an enzyme needed to harden bone. The purpose of this study is to test the safety of the study drug called ENB-0040 and see what effects is has on human juveniles and HPP.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a rare inherited form of rickets and osteomalacia caused by inactivating mutations in the gene encoding the tissue-nonspecific isoenzyme of alkaline phosphatase (TNSALP). The prevalence of the disease is thought to be about 1:100,000 although it is markedly higher in a small Canadian Mennonite population (Fraser 1957, Chodirker 1990). Inheritance can be autosomal recessive or dominant, and penetrance is variable resulting in a wide range of clinical expressivity. HPP differs from other forms of rickets and osteomalacia in that serum levels of calcium and phosphorus are generally normal or even elevated (Whyte 2002). Low circulating levels of alkaline phosphatase with elevated serum or urine levels of the TNSALP substrates inorganic pyrophosphate (PPi), pyridoxal 5'-phosphate (PLP) and phosphoethanolamine (PEA) are the biochemical hallmarks of this inborn error of metabolism.

Disease severity in HPP is inversely related to the age at symptom presentation. The most severe cases occur in utero and almost invariably result in death, generally due to pulmonary compromise. Infants who present in the first six months of life have about 50% mortality. Children and adults have less severe disease but can have frequent fractures, bone pain, bowing of the long bones and muscle weakness, and morbidity is generally cumulative. Some patients cannot ambulate independently and end up wheelchair-bound.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from parent or legal guardian prior to participation
2. Boys >/= 5 and < 12 years of age and girls >/= 5 and < 10 years of age with open growth plates at time of enrollment
3. Documented history of HPP, as evidenced by:

   1. Presence of HPP-related rickets on skeletal radiographs
   2. Serum alkaline phosphatase (ALP) below age-adjusted normal range
   3. Plasma PLP at least twice the upper limit of normal (>/=220 nM)
4. Ambulatory without the use of assistive devices
5. Ability of patient and parent/guardian to comply with study requirements

Exclusion Criteria:

1. Serum calcium or phosphorus below age-adjusted normal range
2. History of sensitivity to any study drug constituent
3. Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities
4. Treatment with an investigational drug within 1 month before start of study drug
5. Current enrollment in any other study involving an investigational new drug, device, or treatment for HPP (eg, bone marrow transplantation)
6. Current evidence of a treatable form of rickets
7. Prior treatment with bisphosphonates
8. Bone fracture or orthopedic surgery within the past 12 months
9. Major congenital abnormality other than those associated with HPP

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Skeletal radiographs using a qualitative Clinical Global Impression of Change (CGI-C) scoring system | 6 months

SECONDARY OUTCOMES:
PK using serum peak and trough levels and PD of plasma inorganic pyrophosphate (PPi) and plasma pyridoxal-5' phosphate (PLP) as biomarkers for HPP. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Whyte, MD, Principal Investigator — Shriners Hospital, St. Louis. MO

REFERENCES:
- [Background] Millan JL, Narisawa S, Lemire I, Loisel TP, Boileau G, Leonard P, Gramatikova S, Terkeltaub R, Camacho NP, McKee MD, Crine P, Whyte MP. Enzyme replacement therapy for murine hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):777-87. doi: 10.1359/jbmr.071213. PMID 18086009
- [Background] Drake MT, Khosla S. Bone-targeted replacement therapy for hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):775-6. doi: 10.1359/jbmr.080305. No abstract available. PMID 18318644